CLINICAL TRIAL: NCT02628015
Title: Theory of Mind Bei Ehemals früh- Und Reifgeborenen Vorschulkindern, Schulkindern, Jugendlichen Und Erwachsenen
Brief Title: Theory of Mind in Preschool Children, School Children, Youths and Adults Born Preterm or Full-term
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Stephanie Braun, Master of Science, Psychologist, University of Bonn
Other Study IDs: ToM-2016-2018
Record Dates: First submitted 2015-11-14; First posted 2015-12-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Premature Birth
Keywords: Theory of Mind; Very Low Birthweight Infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- preschool children preterm: born 2010 or 2011 Birthweight <1500g
- preschool children full-term: born 2010 or 2011 born after 38 weeks
- school children preterm: same children from the preschool group will be tested 2 years later again
- school children full-term: same children from the preschool group will be tested 2 years later again
- youths preterm: born 2001 or 2002 Birthweight <1500g
- youths full-term: born 2001 or 2002 born after 38 weeks
- adults preterm: Birthweight <1500g
- adults full-term: born after 38 weeks

SUMMARY:
This study tests preschoolers, school children, youths and young adults, who were born preterm or full-term, in their theory of mind abilities.

DETAILED DESCRIPTION:
Is there any difference in the development of theory of mind between preterms and full-terms? Is there a risk group of preterms to develop a deficit in theroy of mind?

Four groups are tested: prescoolers (again two years later), youths and young adults.

All participants were tested for theory of mind, executive functions, language and cognitive abilites.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* preterm: birthweight <1500g
* full-term: born after 38 weeks

Exclusion Criteria:

* no informed consent

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: preterms were born in the University Hospital of Cologne
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
theory of mind 1 | up to 7 months
  Theory of Mind Scale (Group 1 and 2)
executive function 1 | up to 7 months
  Teddy-bear-Set-Shifting Task (all groups)
executive function 2 | up to 7 months
  Tower of London (all groups)
Language 1 | up to 7 months
  SETK 3-5 - Language Understanding Task (Group 1)
  there will be only one score for each participant, but there is a different task for the first group, than for the others
cognitive abilities 1 | up to 7 months
  SON 2 1/2 - 7 - Two subtests: Analogies and Categories (group 1) there will be two test-scores for each participant, but they can be aggregated to one score for cognitive abilities
theory of mind 2 | up to 7 months
  Mental State Stories (Group 2, 3 and 4)
theory of mind 3 | up to 7 months
  Faux Pas Stories (Group 2, 3, and 4)
theory of mind 4 | up to 7 months
  Reading the mind in the Eyes Test Revised (Group 4)
theory of mind 5 | up to 7 months
  Cambridge Mindreading Face-Voice Battery (only visual Items) (Group 4)
Language 2 | up to 7 months
  CFT 20 R - Vocabulary Task (group 2,3,4)
cognitive abilities 2 | up to 7 months
  SON 6-40 - Two subtests: Analogies and Categories (group 2,3,4) there will be two test-scores for each participant, but they can be aggregated to one score for cognitive abilities

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Bonn, Germany